CLINICAL TRIAL: NCT04259632
Title: Prolonged Daily Fasting as a Viable Alternative to Caloric Restriction in At-Risk Obese Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MED-2019-28331; R01DK124484 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time Restricted Eating (TRE) (Experimental): For the TRE group, we will restrict the eating window to 8 hours, where they will eat ad libitum. This is the same interval established by Dr. Panda and by our preliminary data. This interval will be entered into the mCC app and participants will be asked to adhere to this eating window during the intervention. All eating occasions will be logged using the mCC app. Only water and medications will be allowed outside of the eating window.
  Interventions: Behavioral: Time Restricted Eating (TRE)
- Caloric Restriction (CR) (Active Comparator): Participants randomized to CR will meet with the study dietitian prior to the intervention and be counseled on options to reduce their caloric intake by 15%, while maintaining their eating window. The 15% reduction was selected as our preliminary data and recent literature suggest that TRE with ad libitum intake reduces caloric intake by ~270 to 300 cal/day. The 15% CR is similar to the 11.9% CR achieved by the CALERIE-2 study, which is a 2 year study of CR.26 All eating occasions will be logged using the mCC app. The weekly dietitian review of the mCC information will include maintenance of the eating window and examination of dietary intake to determine compliance with the 15% CR.
  Interventions: Behavioral: Caloric Restriction (CR)
- Unrestricted Eating (non-TRE) (No Intervention): For the unrestricted eating (non-TRE) group, participants will eat ad libitum per their usual habits. They will receive initial counseling about mCC logging. All eating occasions will be logged using the mCC app.

INTERVENTIONS:
Behavioral: Time Restricted Eating (TRE) — daily eating window restricted to 8 hours
  Arms: Time Restricted Eating (TRE)
Behavioral: Caloric Restriction (CR) — 15% daily caloric deficient
  Arms: Caloric Restriction (CR)

SUMMARY:
Purpose: Obesity is reaching epidemic proportions, affecting 36% of the adult population in the United States. There is intense interest in dietary management to treat obesity and its associated complications. The first line of obesity treatment is caloric restriction (CR), although recidivism is common. For moderate CR, attrition rates of 20% are often reported, therefore weight loss options beyond CR are urgently needed.

DETAILED DESCRIPTION:
Aim#1: Evaluate the effect of TRE with ad libitum intake on weight and body composition.

H 1.1: Individuals in the TRE and CR groups will have similar weight loss, which will be greater than weight loss achieved in the non-TRE group (primary outcome).

H 1.2: TRE will result in greater loss of loss of total body fat (quantified by DXA) and greater loss of hepatic/visceral fat/ectopic fat (quantified by MRI) than CR.

Aim#2: Assess the effect of TRE with ad libitum intake on caloric balance. H 2.1: TRE will reduce caloric intake compared with non-TRE [gold-standard interviewer administered 24-hour dietary recall (primary outcome)] with similar reduction as with CR, H.2.2: Compared with non-TRE, TRE will result in selection of more nutrient dense foods during a supervised meal within their eating window; this selection will be similar to CR. H 2.3 TRE will not alter physical activity, but will increase fat oxidation compared with CR and non-TRE.

Aim#3: Assess the effect of TRE with ad libitum intake on metabolic flexibility.

H 3.1: TRE will enhance metabolic flexibility compared with CR and non-TRE as measured by indirect calorimetry [RQ:Respiratory quotient before and during 2 step 6,6-2H2 hyperinsulinemic-euglycemic clamp: primary outcome].

H 3.2: TRE will improve insulin sensitivity compared with non-TRE and similar to CR.

H 3.3: TRE will augment greater fasting lipolysis compared to CR and non-TRE as measured by [U-13C] palmitate and enhance lipolysis suppression during the 2 step 6,6-2H2 hyperinsulinemic-euglycemic clamp.

If these hypotheses are confirmed, this project has significant impact. First, it will advance understanding of the mechanisms underpinning this innovative intervention. Second, TRE can be a practical means of implementing prolonged fasting on a large scale, thereby transforming the treatment of obesity.

Research reported in this publication was supported by the National Center for Advancing Translational Sciences of the National Institutes of Health Award Number UL1-TR002494. The content is solely the responsibility of the authors and does not necessarily represent the official views of the National Institutes of Health.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30 and ≤ 55 kg/m^2
* Own a smartphone compatible with the myCircadianClock (mCC) phone application
* Self-reported habitual wakening between 5-9 am
* Self reported sleep duration of 6-9 hours
* Weight must be stable [+/- 5 pounds] for at least 3 months prior to the study
* Eating window (time between 1st food intake and last food take) ≥14 hours using mCC
* Insulin resistance based on HOMA-IR≥ 2.5 from screening visit results
* Able to understand English

Exclusion Criteria:

* Use of beta-blockers or medications known to affect weight, such as thiazolidinedione (TZD), insulin, glucagon-like peptide (GLP)-1 agonists, phentermine, or sibutamine
* Shift work (i.e. working from 11pm to 7am)
* Clinically significant medical issues (diabetes, cardiovascular disease, uncontrolled pulmonary disease)
* A history of abnormal laboratory results, such as hematologic (platelets < 100), hepatic (LFTs > 2X nl), renal (Cr > 1.5)
* MRI contraindication (metal in body, claustrophobia)
* Eating window < 12 hours per day
* Unable to consistently document food intake using the mCC app (need at least 2 eating occasions> 6 hours apart on a given day for at least 50% of days)
* Pregnancy
* Illiteracy
* Concern for active eating disorder per screening questionnaire
* Self-reported eating disorder or history of eating disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2025-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Chen DA, Pena RH, Oldenburg N, Wang Q, Helgeson E, Yentzer B, Taddese A, LaPage N, Manoogian ENC, Panda S, Chow LS. Post-intervention sustainability of time-restricted eating versus caloric restriction: a secondary analysis. Int J Obes (Lond). 2025 Nov 28. doi: 10.1038/s41366-025-01968-2. Online ahead of print. PMID 41315749

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Time Restricted Eating (TRE) | Caloric Restriction (CR) | Unrestricted Eating (Non-TRE)
Started | 30 | 29 | 29
Completed | 29 | 26 | 26
Not Completed | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Time Restricted Eating (TRE) | Caloric Restriction (CR) | Unrestricted Eating (Non-TRE) | Total
Number analyzed (Participants) | 30 | 29 | 29 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 29 | 88
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 16 | 48
  Male | 13 | 14 | 13 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 0 | 1 | 3
  White | 23 | 26 | 25 | 74
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Weight will be measured by standard scale and reported in kilograms. This between 2 time points - baseline and 12 weeks
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: Kg
Arm/Group | Time Restricted Eating (TRE) | Caloric Restriction (CR) | Unrestricted Eating (Non-TRE)
Number analyzed (Participants) | 29 | 26 | 26
Kg | -3 [-4.1 to -1.9] | -3.5 [-4.7 to -2.3] | -1.3 [-2.5 to -0.1]

2. Secondary Outcome: Change in Whole Body Percent Fat
Description: Body composition will be measured by dual energy x-ray absorptometry (DXA). Parameters of body composition will be calculated by integrated DXA software. Whole body percent fat will be reported as a percentage.
Time Frame: Baseline, 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change in Visceral Fat
Description: Body composition will be measured by dual energy x-ray absorptometry (DXA). Parameters of body composition will be calculated by integrated DXA software. Visceral fat will be reported in grams.
Time Frame: Baseline, 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change in Lean Mass
Description: Body composition will be measured by dual energy x-ray absorptometry (DXA). Parameters of body composition will be calculated by integrated DXA software. Lean mass will be reported in kilograms.
Time Frame: Baseline, 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change in Fat Mass
Description: Body composition will be measured by dual energy x-ray absorptometry (DXA). Parameters of body composition will be calculated by integrated DXA software. Fat mass will be reported in kilograms.
Time Frame: Baseline, 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change in Caloric Intake
Description: Two interviewer-administered 24-hour dietary recalls will be collected from each participant at baseline and 12 weeks. The recalls will be conducted over the telephone and will be unannounced to minimize measurement reactivity. Diet data will be collected using the Nutrition Data System for Research (NDSR) to calculate Calories. Calories will be averaged across the 2 recalls at each time point. Outcome will be reported as difference between average caloric intake at baseline and 12 weeks. Outcome will be reported in kilocalories (Calories).
Time Frame: Baseline, 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change in Metabolic Flexibility
Description: indirect calorimetry to measure glucose and fat oxidation for ~ 30 minutes before and at the end of the 2 step 4-hour hyperinsulinemic-euglycemic clamp [low-dose (10 mU/m2/min) insulin infusion for 2 hours, high-dose (40 mU/m2/min) insulin infusion for 2 hours] Fluctuations in VO2 and VCO2 in the first 5-10 minutes of data acquisition were removed and the mean VO2 and VCO2 at steady state was used for data analysis. The respiratory exchange ratio (RER) was calculated by VCO2 / VO2. . Metabolic flexibility was calculated by the RERclamp-RERrest
Time Frame: baseline, 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Time Restricted Eating (TRE) | Caloric Restriction (CR) | Unrestricted Eating (Non-TRE)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 1/30 | 1/29 | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Time Restricted Eating (TRE) (N=30) | Caloric Restriction (CR) (N=29) | Unrestricted Eating (Non-TRE) (N=29)
ER eval for TIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
ER evaluation for kidney stones and diverticulosis (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT04259632/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT04259632/SAP_001.pdf
  • Informed Consent Form (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT04259632/ICF_002.pdf